CLINICAL TRIAL: NCT03486496
Title: An Open-label Phase II Trial of Gefitinib and Berberine in Patients With Advanced Non-small Cell Lung Cancer and Activating EGFR Mutations
Brief Title: Gefitinib and Berberine in the First-line Treatment of Lung Adenocarcinoma With EGFR Mutation
Acronym: Geber
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSWOF201801
Record Dates: First submitted 2018-03-24; First posted 2018-04-03 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Lung Adenocarcinoma; EGFR Mutation
Keywords: Lung Adenocarcinoma; EGFR mutation; Gefitinib; Berberine
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — Gefitinib; Berberine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gefitinib and Berberine (Experimental): Experimental: Gefitinib and Berberine Patients will be treated with Gefitinib and Berberine. Gefitinib: 250 mg p.o., daily. Berberine: 50 mg p.o., tid.
  Interventions: Drug: gefitinib; Drug: Berberine

INTERVENTIONS:
Drug: gefitinib — Patients will be treated with gefitinib, 250 mg p.o., daily
  Other Names: Iressa (AstraZeneca)
Drug: Berberine — Patients will be treated with Berberine, 50 mg p.o., tid
  Other Names: Berberine Sulfate

SUMMARY:
Rationale:

Advanced non-small-cell lung cancer (NSCLC) patients harboring epidermal growth factor receptor (EGFR) mutations (del19 or L858R) show an impressive progression-free survival between 9 and 11 months when treated with gefitinib. Combination of gefitinib and berberine could improve efficacy in lung cancer with EGFR mutation in vivo and vitro. The investigators hypothesize that progression-free survival could be improved by combination of gefitinib and berberine.

DETAILED DESCRIPTION:
Strong lipogenic activity and high expression of sterol regulatory element-binding protein 1 (SREBP-1) were found in gefitinib-resistance NSCLC cells. Berberine, an effective suppressor of SREBP1 and lipogenesis regulated through ROS/AMPK pathway, selectively inhibited the growth of gefitinib-resistance NSCLC cells but not that of normal cells. It effectively caused mitochondrial dysfunction, activated reactive oxygen species (ROS)/AMPK pathway and finally suppressed cellular lipogenesis and cell proliferation. Addition of ROS blocker, AMPK inhibitor and palmitic acid significantly reduced the effect of Berberine. In in vivo study, treatment of Berberine led to significant inhibition of mouse tumor xenograft growth.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ECOG performance status 0-2
* Adequate haematological function, coagulation, liver function and renal function
* Pathological diagnosis of predominantly non-squamous, non-small-cell lung cancer (NSCLC)
* TNM version 7 stage IV disease including M1a (malignant effusion) or M1b (distant metastasis), or locally advanced disease not amenable to curative treatment (including patients progressing after radiochemotherapy for stage III disease)
* Measurable or evaluable disease (according to RECIST 1.1 criteria).
* Centrally confirmed EGFR exon 19 deletion (del19) or exon 21 mutation (L858R)

Exclusion Criteria:

* Patients who have had in the past 5 years any previous or concomitant malignancy EXCEPT adequately treated basal or squamous cell carcinoma of the skin, in situ carcinoma of the cervix or bladder, in situ breast carcinoma.

Patients with any known significant ophthalmologic anomaly of the ocular surface

* Patients who received prior chemotherapy for metastatic disease
* Patients who received previous treatment for lung cancer with drugs targeting EGFR or VEGF
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-06-05 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Within 6 months of the last visit of last patient, approximately 30 months after inclusion of first patient
  Time from the date of enrolment to discontinuation of treatment for any reason (including progression of disease, treatment toxicity, refusal and death)

SECONDARY OUTCOMES:
Objective response | through study completion,an average of three years
  Best overall response (complete remission or partial remission) across all assessment time-points according to RECIST Criteria 1.1, during the period from enrolment to termination of trial treatment.
safety | Within 6 months of the last visit of last patient, approximately 30 months after inclusion of first patient
  Adverse events graded according to NCI CTCAE V4.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Huang, MD., Principal Investigator — Fujian Cancer Hospital
Locations (1):
- Fujian cancer hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data access requests will be reviewed by an external indepentent Review Panel. Requesdtors will be required to sign a Data Access Agreement.

REFERENCES:
- [Result] Fan XX, Leung EL, Xie Y, Liu ZQ, Zheng YF, Yao XJ, Lu LL, Wu JL, He JX, Yuan ZW, Fu J, Wei CL, Huang J, Xiao DK, Luo LX, Jiang ZB, Zhou YL, Kam RK, Liu L. Suppression of Lipogenesis via Reactive Oxygen Species-AMPK Signaling for Treating Malignant and Proliferative Diseases. Antioxid Redox Signal. 2018 Feb 10;28(5):339-357. doi: 10.1089/ars.2017.7090. Epub 2017 Aug 4. PMID 28665143